CLINICAL TRIAL: NCT03437928
Title: Deep Brain Stimulation (DBS) for Depression Using Directional Current Steering and Individualized Network Targeting
Brief Title: DBS for Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Texas (Other)
Responsible Party: Principal Investigator, Sameer Sheth, Professor, Vice-Chair of Clinical Research, Department of Neurosurgery, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-43036; NCT03964194 (obsolete NCT alias)
Record Dates: First submitted 2018-01-09; First posted 2018-02-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder (MDD); MDD; Neuromodulation; Deep Brain Stimulation (DBS); DBS; Electrophysiology; Imaging
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Directional Deep Brain Stimulation (Experimental)
  Interventions: Device: Directional Deep Brain Stimulation

INTERVENTIONS:
Device: Directional Deep Brain Stimulation — Boston Scientific Vercise DBS leads and 16-channel implanted pulse generators (IPGs) will be implanted to control the shape and size of stimulation

SUMMARY:
The goal of the study is to address the unmet need of TRD patients by identifying brain networks critical for treating depression and to use next generation precision DBS with steering capability to engage these targeted networks. The study's goal will be achieved through 3 specific aims:

1. Demonstrate device capability to selectively and predictably engage distinct brain networks
2. Delineate depression-relevant networks and demonstrate behavioral changes with network-targeted stimulation
3. Demonstrate that chronic DBS using steered, individualized targeting is feasible and safe for reducing depressive symptoms

DETAILED DESCRIPTION:
Treatment-resistant depression (TRD) is a major worldwide burden. Major depression has a lifetime prevalence of ~15% across developed countries. Up to a third of patients fail to respond adequately to evidence-based treatments, including pharmacological, behavioral, and electroconvulsive therapy. The investigators employ an innovative approach, including subacute invasive neurophysiological monitoring with which they aim to gain insight into the networks underlying depression symptomatology, confirm the ability to predict the effects of precision DBS on network activity, and harmonize these insights to implement network-guided DBS for TRD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) between ages 22 and 70;
2. DSM-5 diagnosis (assessed by Structured Clinical Interview for DSM-5 Axis I disorders SCID-5) of major depression disorder (MDD) as the primary diagnosis. A current major depressive episode (MDE), recurrent or single episode with first episode before age 60, secondary to nonpsychotic unipolar major depressive disorder;
3. Chronic illness with current MDE ≥24 months duration and/or recurrent illness with at least a total of 2 lifetime episodes (including current episode >12 months);
4. Treatment resistance (defined by criteria on the Antidepressant Treatment History Form ATHF): Failure (i.e. persistence of the major depressive episode) to respond to a minimum of four adequate depression treatments from at least two different treatment categories (e.g. SSRIs, SNRIs, TCAs, other antidepressants, lithium-addition, irreversible MAOIs, antidepressant augmentation with an atypical antipsychotic medication);
5. Previous trial of Electroconvulsive Therapy (ECT) (lifetime): either did not respond, relapsed, poorly tolerated or refused. If refused, will discuss reasons and ensure subject understands relative risks of ECT versus DBS. We will try to enrich sample with patients who had previously shown response to ECT (or another intervention) that was partial or un-sustained;
6. Symptom severity for Screening: Hamilton Depression Rating Scale-17 item (HDRS17) ≥20;
7. The HDRS17 must remain greater than or equal to 20 on two separate assessments (at initial screening and 1 week before surgery), over a 1-month period;
8. Symptom severity for Outcome: Montgomery Asberg Rating Scale (MADRS) ≥27 to be met at assessment one-week pre-op;
9. Lifetime exposure to minimal 6 weeks of psychotherapy without sustained response;
10. Must have a brain MRI within 3 months of enrollment that is "normal", according to the radiology report, or does not reveal any findings that in the opinion of the Investigator preclude participation in the study;
11. Stable antidepressant medication regimen for the month preceding surgery;
12. Modified mini-mental state examination (MMSE) score ≥ 24;
13. Normal thyroid stimulating hormone (TSH) level within 12 months of study entry;
14. The patient does not have any medical or physical conditions which, in the opinion of the Investigator, make it unlikely the patient will be able to participate for the duration of the study;
15. Able and willing to give informed consent and agree to attend regular clinic visits for at least 12 months following surgery;
16. Must have a treating psychiatrist, a family member, significant other/living partner, a caregiver, or a person known by the subject present at the Screening visit for the discussion about the study before co-signing the informed consent form;
17. Willingness to sign Treatment Contract;
18. Agrees to be followed at regular intervals by a licensed psychiatrist and to provide written permission allowing any and all forms of communication between the research team and the subject's healthcare providers, for the entirety of the study.

Exclusion Criteria:

1. DSM-5 Axis I Disorders: any lifetime history of psychotic disorder (e.g., schizophrenia, schizoaffective disorder);
2. Bipolar disorder with rapid cycling and history of manic episode requiring hospitalization within the past 5 years;
3. Clinically significant Cluster A or B personality disorder;
4. Alcohol or substance use disorder within 6 months, excluding nicotine;
5. Urine drug test positive for illicit drugs;
6. Any evidence or indication of suicidal intent, suicidal attempt, or suicidal behavior, including but not limited to the C-SSRS score, within the past one year;
7. Neurological/Medical condition that makes the patient, in the opinion of the surgeon, a poor surgical candidate (e.g., progressive neurodegenerative disorder, significant cardiopulmonary disorder, need for chronic anticoagulation);
8. Any history of seizure disorder, hemorrhagic stroke, or has high risk of seizure (history of congenital malformation, history of brain injury, neuro-developmental disorder, currently taking medication that is known to lower seizure threshold, or other factors that predispose seizures);
9. Any medical contraindication to surgery such as infection;
10. Coagulopathy: Bleeding propensity and/or one of the following: INR > 1.5; prolonged activated partial thromboplastin time (aPTT) ≥ 45 sec; platelet count < 100×103/uL;
11. A blood pressure of ≥ 180/110 mmHg at a single visit and evidence of cardiovascular disease (CVD);
12. Participation in another drug, device, or biological trial within 90 days;
13. Current implanted stimulation devices including cardiac pacemakers, defibrillators, and neurostimulators including spinal cord stimulators and deep brain stimulators;
14. Pregnant or has plans to become pregnant in the next 24 months;
15. Anticipated need for MRI;
16. Need for Diathermy;
17. Chronic use of anticoagulant or anti-platelet agents that cannot be safely stopped for a sufficient duration (minimum 2.5 weeks) in the peri-operative period;
18. Any Psychiatric/Neurological/Medical condition that makes the subject, in the opinion of the Investigator, a poor candidate.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms | 54 to 60 months
  Response will be defined as 50% decrease in Montgomery-Asberg Depression Rating Scale (MADRS) from baseline. The range is from 0 to 60 and a score higher than 20 indicates moderate to severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer A Sheth, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Noecker AM, Mlakar J, Bijanki KR, Griswold MA, Pouratian N, Sheth SA, McIntyre CC. Stereo-EEG-guided network modulation for psychiatric disorders: Interactive holographic planning. Brain Stimul. 2023 Nov-Dec;16(6):1799-1805. doi: 10.1016/j.brs.2023.11.003. Epub 2023 Dec 20. PMID 38135359
- [Derived] Powell MP, Anso J, Gilron R, Provenza NR, Allawala AB, Sliva DD, Bijanki KR, Oswalt D, Adkinson J, Pouratian N, Sheth SA, Goodman WK, Jones SR, Starr PA, Borton DA. NeuroDAC: an open-source arbitrary biosignal waveform generator. J Neural Eng. 2021 Feb 5;18(1):10.1088/1741-2552/abc7f0. doi: 10.1088/1741-2552/abc7f0. PMID 33152715